CLINICAL TRIAL: NCT04335864
Title: A Clinical Trial Comparing Laparoscopic Salpingectomy Versus Hysteroscopic Proximal Tubal Occlusion on Pregnancy Rates Following ICSI (Intra-Cytoplasmic Sperm Injection) in Infertile Cases of Hydrosalpinx.
Brief Title: Comparing the Impact of 2 Different Techniques in Management of Hydrosalpinx on Pregnancy Rates Following ICSI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Shaimaa Mostafa Mohammed Refaay El shemy, Principal investigator, Lecturer in obstetrics and gyneocolgy department, Cairo university, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Hydrosalpinx and ICSI
Record Dates: First submitted 2020-03-29; First posted 2020-04-06 (Actual); Last update posted 2021-06-29 (Actual); Status verified 2021-06

CONDITIONS: Hydrosalpinx

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Active Comparator): 39 patients with hydrosalpinx will have laparoscopic salpingectomy
  Interventions: Procedure: Laparoscopic salpingectomy
- Group B (Active Comparator): 39 patients with hydrosalpinx will have hysteroscopic proximal tubal occlusion
  Interventions: Procedure: Hystroscopic proximal tubal occlusion

INTERVENTIONS:
Procedure: Laparoscopic salpingectomy — 39 patients with hydrosalpinx will have laparoscopic salpingectomy
  Arms: Group A
Procedure: Hystroscopic proximal tubal occlusion — 39 patients with hydrosalpinx will have hysteroscopic proximal tubal occlusion
  Arms: Group B

SUMMARY:
Assessment and comparing pregnancy outcomes in hydrosalpinx patients treated by hysteroscopic tubal occlusion and laparoscopic salpingectomy before ICSI.

DETAILED DESCRIPTION:
Hydrosalpinx has a detrimental effect on the rates of implantation, pregnancy and early pregnancy loss following IVF. A meta-analysis demonstrated that the implantation rate and clinical pregnancy rate decreased by 50% in patients with hydrosalpinx. The negative consequences could be due to embryotoxic properties, a decrease in endometrial receptivity, and hydrosalpinx fluid mechanically flushing the embryo from the uterus.

Although laparoscopic salpingectomy and laparoscopic proximal ligation increase ongoing pregnancy rates in women with hydrosalpinges, those interventions are invasive and carry anaesthetic and surgical risks, especially in the presence of extensive adhesions, often seen in women with hydrosalpinges. In view of the possible adverse effects of laparoscopic surgery, an alternative less-invasive treatment for hydrosalpinges prior to IVF would be useful.

The effectiveness of hysteroscopic tubal occlusion when compared with salpingectomy has not been established. Randomized clinical trials comparing both procedures prior to IVF are lacking.

The present study was designed to compare hysteroscopic tubal occlusion and laparoscopic salpingectomy in the treatment of hydrosalpinges prior to IVF.

This study hypothesized that in women scheduled for IVF/ICSI hysteroscopic proximal occlusion of hydrosalpinges would be non-inferior to laparoscopic salpingectomy in terms of ongoing pregnancy rates following IVF/ICSI.

ELIGIBILITY:
Inclusion Criteria:

* primary or secondary infertility cases
* unilateral or bilateral hydrosalpinx proved by HSG (hystersalpingogram) or by TVUS(transvaginal ultrasound) .

Exclusion Criteria:

* Uterine factor of infertility
* male factor of infertility
* preexisting ovarian pathology
* Presence of septic focus
* medical or surgical conditions that contraindicated pregnancy

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 78 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2020-10-30 (Actual); Study Completion 2020-12-15 (Actual)

PRIMARY OUTCOMES:
Clinical pregnancy rate following ICSI | 14 days after Embryo transfer
  Defined as positive qualitative bhcg(beta human chorionic gonadotropin)

SECONDARY OUTCOMES:
Ongoing pregnancy following ICSI | 8 weeks after Embryo transfer
  Defined as positive fetal heart rate on ultrasound at 8weeks gestation

CONTACTS AND LOCATIONS:
Locations (1):
- Kasr Alainy hospital-cairo University, Cairo, Egypt